CLINICAL TRIAL: NCT00646451
Title: A 17 Week, Investigator-initiated, Single-center, Double-blind, Randomized, Placebo-controlled, Cross-over Trial of Pregabalin in Essential Tremor
Brief Title: Pregabalin in the Treatment of Essential Tremor
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Joseph Jankovic, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-19086
Record Dates: First submitted 2007-12-28; First posted 2008-03-28 (Estimated); Results first posted 2021-03-12 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Essential Tremor
Keywords: Essential tremor; Activities of Daily Living (ADL's)
MeSH Terms: conditions — Essential Tremor | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Lyrica) (Active Comparator): Pregabalin (Lyrica) 75 mg bid to a maximum dose of 300 mg bid
  Interventions: Drug: pregabalin (Lyrica)
- Placebo (Placebo Comparator): Placebo to 4 capsules bid
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pregabalin (Lyrica) — 75 mg bid to 300 mg bid based on per subject tolerability
  Other Names: pregabalin
  Arms: Pregabalin (Lyrica)
Drug: placebo — up to 4 capsules bid as tolerated
  Arms: Placebo

SUMMARY:
Pregabalin is approved for the treatment of nerve pain as well as an additional therapy in the treatment of seizures. In December 2004, Pfizer gained Food and Drug Administration (FDA) approval for use of pregabalin in nerve pain associated with diabetes and shingles; making it the first FDA-approved treatment for both of these nerve pain states.

Tremor is uncontrolled trembling in part of the body. Essential tremor (ET) is associated with purposeful movement(e.g., holding a glass to drink, shaving, writing and buttoning a shirt). It occurs most often in the hands and head and also may affect the arms, voice box (larynx), trunk, and legs. ET is caused by abnormalities in areas of the brain that control movement. It usually does not result in serious complications.

ET affects approximately 5 million people in the United States. Incidence is highest in people over the age of 60.

ET usually develops gradually during middle age or later in life. Symptoms may remain mild or become more severe over time. Stress, fatigue, anxiety, and hot or cold weather can worsen the disorder. Severe tremor may cause difficulty doing activities of daily living, such as:

* Brushing hair and teeth
* Holding a glass without spilling
* Performing self-care (e.g., getting dressed, shaving, putting on makeup)
* Using eating utensils
* Writing and drawing

The purpose of this pilot/feasibility study is to examine the tolerability and efficacy of Pregabalin in patients with ET.

In other words, can patients diagnosed with ET tolerate high dose of pregabalin? Will the pregabalin be considered as an efficient medicine in the treatment of ET?

DETAILED DESCRIPTION:
Overview We propose a single site, double-blind, placebo-controlled, cross-over design. Drug will be administered in 75mg capsules with a target dose of 300 mg/day. Pregabalin will be titrated upward as described in the "Summary of Schedule" table with flexibility. During weeks 3-5 and 12-14, the investigator will have the option of increasing the study drug from 2 capsules per day (150 mg vs. placebo) to 3 or 4 capsules per day if no benefit is noted. If the dose is increased, it must be done so at a rate of 150mg/day/week. Patients who can not tolerate a higher dose will be allowed to drop back to a previously tolerated dose but must be on that dose for one week prior to evaluation. After treatment and clinical assessment, study drug will be decreased by 150mg/day every 2 days until discontinuation. This pertains to both the wash out phase and at the end of the study. Both adverse events and need for drug titration will be conducted during the safety call.

Identical assessments will be done at baseline and at the end of the treatment period for both drug and placebo. Half of the subjects (group A) will initiate with placebo and then crossover to drug. The other half (group B) will start treatment with pregabalin and then crossover to placebo.

The primary endpoint will be the change in Fahn-Tolosa-Marin Tremor Rating Scale (TRS) from baseline. Scale has Parts A= (severity of rest, action & postural tremor in upper and lower extremities, face, voice, tongue, head & trunk), B= (severity of tremor writing, drawing & pouring), C= (functional disability while speaking, eating, drinking, maintaining hygiene, dressing & working) and the total summed.

Other clinical assessments will include Clinical Global Impression of Change (CGI-C), Quality of Life in Essential Tremor Questionnaire (QUEST) maximum score =100, Hamilton Anxiety Scale (HAM-A) score 0-17 = mild, 18-24 = moderate, and 25-30 moderate to severe, and a sleep hygiene questionnaire rating across 5 domains- physical symptoms, energy & motivation, concentration, interpersonal relations, and psychological symptoms (HD-16). For the TRS, HAM-A, QUEST, and HD-16 higher scores represent increased symptom severity or diminished quality of life and the CGI-C is scored as follows: 1=very much improved, 2=much improved, 3= mildly improved, 4=no change, 5= mildly worse, 6= much worse, and 7=very much worse.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be between the ages of 18 and 80 inclusive.
2. Each subject must have current manifestations of ET symptoms based on the Tremor Investigational Group (TRIG) criteria for definite or probable ET: - Moderate or severe tremor in head or arms for at least 3 years duration. - No present causes of enhanced physiologic tremor. - No recent exposure to tremorogenic drugs or drug withdrawal states. - No direct or indirect trauma to the nervous system within 3 months preceding the onset of tremor. - No historic or clinical evidence of psychogenic tremor origin.
3. Subjects with a history of seizures are eligible.
4. Subjects must be in generally good health as evidenced by previous medical history and clinical examination.
5. Patients will be allowed to take Beta-blockers but will not be allowed to take any other medication for tremor (primidone, topiramate, benzodiazepines, etc.) An evening dose of a benzodiazepine to improve sleep is acceptable. They must have been on a stable dose of any existing beta-blocker for 4 weeks prior to entry into the study and will not be allowed to change the dose of that medication throughout the controlled portion of the study. Any medication discontinued during screening in order to comply with these criteria must be stopped for 5 half-lives prior to study initiation.
6. Subjects must be accessible by telephone.
7. If the subject is a female of childbearing age, she must have had a hysterectomy, tubal ligation, otherwise be incapable of pregnancy, or have practiced one of the following methods of contraception for at least one month prior to study entry (or a negative urine pregnancy test within one week of study entry): - Hormonal contraceptives - Spermicide and barrier - Intrauterine device - Partner sterility
8. Prior to participation in this study, each subject must sign an informed consent.

Exclusion Criteria:

1. Patients do not meet TRIG criteria for probable ET.
2. Subjects who are not able to abstain from alcohol for 24 hours prior to each evaluation.
3. Patients who can not maintain an identical dose of any medicine that may affect tremor during their entire study involvement.
4. Subjects who have exhibited any psychotic symptomatology.
5. Subjects who have known renal deficiencies.
6. Subjects who have been intolerant of pregabalin in the past
7. Prior surgical treatment for tremor.
8. Patients currently taking more than a single drug for ET.
9. Patients taking anti-seizure medications.
10. Breast feeding or pregnant females.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Jankovic, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- PDCMDC 6550 Fannin, Suite 1801, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrara JM, Kenney C, Davidson AL, Shinawi L, Kissel AM, Jankovic J. Efficacy and tolerability of pregabalin in essential tremor: a randomized, double-blind, placebo-controlled, crossover trial. J Neurol Sci. 2009 Oct 15;285(1-2):195-7. doi: 10.1016/j.jns.2009.06.044. Epub 2009 Jul 25. PMID 19631949

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin First, Then Placebo: Pregabalin: 75 mg bid to 300 mg bid based on per subject tolerability. Study crossover design. Patients were randomized for treatment with PGB or placebo, titrated over 6 weeks.
- Placebo First, Then Pregabalin: Placebo capsules: up to 4 capsules bid as tolerated. Study crossover design. Patients were randomized for treatment with PGB or placebo, titrated over 6 weeks.
Period: Overall Study
Arm/Group | Pregabalin First, Then Placebo | Placebo First, Then Pregabalin
Started | 10 | 10
Completed | 6 | 10
Not Completed | 4 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Exacerbation of pre-existing condition | 1 | 0

BASELINE CHARACTERISTICS:
Population: Study crossover design. Patients were randomized for treatment with PGB or placebo, titrated over 6 weeks. TRS (primary endpoint), then CGI-C, QUEST, HAM-A, and HD-16 secondary endpoints at end of treatment periods for both drug and placebo.
Groups:
- All Participants: Demographics and clinical characteristics of participants at study initiation are listed in Table 1 of the paper. Sixteen of 20 patients completed the study and were included in the analysis of drug efficacy (Table 2).
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Tremor Rating Scale (TRS) [Mean (Standard Deviation); unit: units on a scale] — a TRS part A rates the severity of resting, postural and action tremor in upper and lower extremities, face, tongue, voice, head and trunk. Part B rates the severity of upper extremity tremor while writing, drawing, and pouring liquid. Part C rates functional disability of tremor while speaking, eating, drinking, maintaining hygiene, dressing, and working. (0: no tremor, 1: barely perceptible tremor, 2: < 2 cm, 3: 2-4 cm, and 4: > 4 cm). The higher scores represent increased symptom severity or diminished QoL.
  units on a scale
    TRS Part A | 18.3 (6.0)
    TRS Part B | 50.8 (16.4)
    TRS Part C | 43.1 (16.3)
    TRS total | 37.1 (11.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Tremor Rating Scale (TRS) Compared With Baseline.
Description: Change from baseline in the overall TRS score obtained at the final evaluation (end of study). The overall TRS score will be derived from the three TRS subscales. The minimum and maximum score for part A is 0-80, part B is 0-36, and part C is 0-28 giving a maximum score of 144. TRS part A rates the severity of resting, postural and action tremor in upper and lower extremities, face, tongue, voice, head and trunk. Part B rates the severity of upper extremity tremor while writing, drawing, and pouring liquid. Part C rates functional disability of tremor while speaking, eating, drinking, maintaining hygiene, dressing, and working. Higher scores represent increased symptom severity or diminished quality of life.
  .
Time Frame: baseline to 6 weeks
Population: Indistinguishable capsules and an identical titration protocol were used for PGB and placebo. Patients received the study drug at an initial dose of 75 mg twice daily, with upward titration to a target dose of 150 mg bid up to 300 mg bid. The study drug was increased at a rate of 150 mg/day/week.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 1-Pregabalin: pregabalin : 75 mg bid to 300 mg bid based on per subject tolerability. Crossover study design and measure change in TRS Pregabalin group versus placebo group.
- 2-Placebo: placebo capsules : up to 4 capsules bid as tolerated. Crossover study design and measure change in TRS Pregabalin group versus placebo group.
Arm/Group | 1-Pregabalin | 2-Placebo
Number analyzed (Participants) | 20 | 16
units on a scale
  TRS Part A | 2.4 (4.7) | -0.2 (4.1)
  TRS Part B | 6.7 (12.3) | 3.6 (6.6)
  TRS Part C | 4.5 (13.9) | -1.5 (12.8)
  Total TRS | 5.1 (9.7) | 0.3 (4.6)

2. Secondary Outcome: Secondary Outcome Measures Quality of Life in Essential Tremor (QUEST), Hamilton Anxiety Scale (HAM-A), Hotel Dieu-16 a Sleep Hygiene Questionnaire(HD-16), and Clinical Clobal Impression-Change Scale (CGI-C)
Description: The Quality of Life in Essential Tremor Questionnaire (QUEST), Hamilton Anxiety scale (HAM-A) and Hotel Dieu-16 (HD-16) were scored as per published guidelines [7], [8] and [9]. The QUEST rates patient perception as influenced by tremor across 5 domains. A QUEST score will be between 0 and 120 with 0 = no essential tremor and 120 = severe essential tremor. The HAM-A rates the severity of anxiety symptomatology across 14 parameters. Scores of 14-17 = mild anxiety, 18-24 = moderate anxiety, and 25-30 = severe anxiety; The HD-16 rates insomnia-related quality of life across five domains. An HD-16 score of 73.1 - 248.5 = severe insomnia, 61-73.1 = mild insomnia, and 0 - 61 = good sleeper. For the scales, HAM-A, QUEST and HD-16, higher scores represent increased symptom severity or diminished quality of life. CGI-C was scored as follows: 1 = very much improved, 2=much improved, 3=mildly improved, 4=no change, 5=mildly worse, 6= much worse, and 7= very much worse.
Time Frame: baseline to 6 weeks
Population: Change in secondary measures of efficacy compared with baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pregabalin: Patients received the study drug at an initial dose of 75 mg twice daily, with upward titration to a target dose of 150 mg twice daily. Patients were given the option to increase the study drug to as high as 300 mg twice daily if inadequate benefit was perceived after 3 weeks of treatment. The study drug was increased at a rate of 150 mg/day/week. All patients in both periods were contacted by phone after two weeks of treatment to facilitate drug titration and address any adverse events. Patients were permitted to return to a lower dose if side effects occurred during drug titration.
  After assessment protocols were completed, patients were titrated off the study drug at a rate of 150 mg every 2 days until discontinuation.
- Placebo: Patients received the study drug/matching placebo at an initial dose of 75 mg twice daily, with upward titration to a target dose of 150 mg twice daily. Patients were given the option to increase the study drug to as high as 300 mg twice daily if inadequate benefit was perceived after 3 weeks of treatment. The study drug was increased at a rate of 150 mg/day/week. All patients in both periods were contacted by phone after two weeks of treatment to facilitate drug titration and address any adverse events. Patients were permitted to return to a lower dose if side effects occurred during drug titration.
  After assessment protocols were completed, patients were titrated off the study drug at a rate of 150 mg every 2 days until discontinuation.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 20 | 16
units on a scale
  QUEST | 8.0 (20.3) | -9.7 (14.5)
  HAM-A | 1.1 (5.2) | 4.1 (5.4)
  HD-16 | 32.2 (146.8) | -38.6 (99.3)
  CGI-C | 3.9 (1.3) | 3.8 (0.5)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Outcome on study completers was assessed via ANOVA models using a 2 × 2 Latin-square crossover design including sequence, period, and treatment effects. A significant carryover effect was excluded. Analyses were performed using Stata IC version 10.0 for Windows. Unfortunately the small sample size of our study limits the possibility of a meaningful post-hoc analysis targeted to these variables; Test type: Superiority or Other; p = 0.162, ANOVA; The Quest rates patient perception of health status as influenced by tremor across 5 domains, physical, psychosocial, communication, hobbies/leisure, and work/finance. HAM-A rates severity of anxiety symptomatology across 14 parameters. Scores of 14-17 correspond to mild anxiety, scores of 18-24 is moderate anxiety and 25-30 severe anxiety. HD-16 rates insomnia-related QoL across 5 domains: physical symptoms, energy & motivation, concentration, interpersonal relations and psychological symptoms. These scales were scored per published guidelines

ADVERSE EVENTS:
Time Frame: 14 weeks of study duration
Groups:
- Pregabalin: pregabalin: 75 mg bid to 300 mg bid based on per subject tolerability
- Placebo: placebo capsules: up to 4 capsules bid as tolerated
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 14/20 | 9/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=20) | Placebo (N=18)
drowsiness (General disorders) | 5 (5) | 3 (3)
dizziness (General disorders) | 4 (4) | 1 (1)
fatigue (General disorders) | 3 (3) | 0 (0)
instability (General disorders) | 3 (3) | 1 (1)
insomnia (General disorders) | 0 (0) | 2 (2)
headache (General disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
This is a investigator initiated trial that was completed in 2008 under 42 CFR 11.22 (b) and does not meet criteria. The study was a pilot and did not lead to registration nor to indication so this level of reporting is not be warranted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No